CLINICAL TRIAL: NCT03752567
Title: "The Community Pharmacist and the Case Management of Diabetic Patient" - No Profit Observational Study on the Role of the Community Pharmacist and the "Pharmacy of the Services" in the Diabetic Patient Case Management
Brief Title: New Patient Support Program in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Farmacia La Regina s.r.l. (Other)
Collaborators: Federfarma Campania (Other); Federfarma Salerno (Other); Health Telematic Network (Industry); Biochemical Systems International S.p.A. (Industry); Next Sight srl (Industry)
Responsible Party: Principal Investigator, Raffaele La Regina, Community pharmacist, Farmacia La Regina s.r.l.
Other Study IDs: 1
Record Dates: First submitted 2018-11-09; First posted 2018-11-26 (Actual); Results first posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: adherence; terapy; follow up; community pharmacy; pharmacist; case manager; telemedicine; pharmacy of service; fundus camera; ecg; local pharmacist; general physician
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group study: Follow up of the patients for 12 months by the community pharmacist in the role of case manager and execution of the activities foreseen by the PAI (individual assistance plan) through telemedicine (ecg, fundus oculi, ankle arm index) and self analysis (glycated hemoglobin, lipid profile, uric acid microalbuminuria).
  Interventions: Other: Follow up

INTERVENTIONS:
Other: Follow up — like group descriptions

SUMMARY:
Non-profit observational study on the role of the community pharmacist and the "pharmacy of services" in the case management of the diabetic patient

DETAILED DESCRIPTION:
Over the last few years, the Italian National Health Service has witnessed numerous and substantial changes, even more evident if one looks at the workload that this system is called to face when it comes to chronic diseases. In fact, while the progress of science has led to better outcomes in the treatment of acute diseases resulting in an increase in the average age of the population and an increase in the number of people suffering from chronic diseases, even multiple, on the other the changed socio-economic conditions activities have led to an increase in the number of elderly and socially fragile individuals. It takes very little to understand that these epidemiological and socio-sanitary mutations pose a serious threat to the stability of the investigator's health system.

To meet these new needs, the different countries of the world are analyzing and adopting various models of chronic disease management. Even if with different methodologies, all the models developed so far put the patient at the center of attention, in its uniqueness and with its needs, and propose to provide the latter with complete assistance, through the integration of health and social services.

In this scenario, also the role of pharmacist, historically linked to the dispensation of drugs upon presentation of a medical prescription and to a final control action to ensure a delivery of medicines in total safety, over time has evolved. In order to carry on this evolution, the pharmacist has been asked for new skills, to realize what has been defined as "the pharmacy of services", through which the pharmacist is recognized the possibility of becoming a strategic figure to meet the changed needs of the population on the one hand and the Italian National Health System on the other and to support the latter in the transition from a "waiting" medicine to an "initiative" medicine.

Diabetic disease and the resulting chronic complications, today, have a very significant impact on patients and their families, on morbidity and mortality, as well as having a strong economic impact on the health system. Despite this, most of the patients do not carry out what is foreseen by their diagnostic therapeutic assistance path (PDTA) due to several reasons such as long waiting times, the need to move to undergo examinations, which is not so easy for young people of working age as well as older people, lack of homogeneity in access to care and in the provision of services and more. The community pharmacist, therefore, represents, for the position in which it is located within the Italian National Health Service, a potential not yet considered. In fact, it could take on the role of case manager (a professional who manages one or more cases entrusted to him according to a pre-established path, such as PDTA, in a defined space-time context) of the patient suffering from type 2 diabetes mellitus due to the capillarity territory, to the hourly availability superior to any other territorial health structure, to the health skills in its possession and to what it can offer in terms of services within the so-called "pharmacy of service".

In this scenario, the pharmacist would not replace any of the other actors already present in the multidisciplinary care team but would integrate in the same and, moreover, being already an agreement with the Italian National Health Service, the conferral of this role would not cause a excessive increase in costs, such as that resulting from the hiring of new staff to achieve the same objectives.

ELIGIBILITY:
Criteria Inclusion:

* age> 18 years,
* patients with type 2 diabetes mellitus diagnosis;
* able to express consent to the study.

Exclusion Criteria:

- Nobody

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with type 2 diabetes mellitus
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele La Regina, dr, Principal Investigator — Farmacia La Regina s.r.l.
Locations (1):
- Farmacia La Regina dott. Rocco Vito, San Rufo, Salerno, Italy

IPD SHARING:
Plan to Share IPD: No
The data will be shared only in aggregate and anonymous form.

REFERENCES:
- [Background] Gerber BS, Rapacki L, Castillo A, Tilton J, Touchette DR, Mihailescu D, Berbaum ML, Sharp LK. Design of a trial to evaluate the impact of clinical pharmacists and community health promoters working with African-Americans and Latinos with diabetes. BMC Public Health. 2012 Oct 23;12:891. doi: 10.1186/1471-2458-12-891. PMID 23088168
- [Background] Brophy L, Williams A, Berman EJ, Keleti D, Michael KE, Shepherd M, Fox SA, Jacobs C, Tan-Torres S, Gelzer AD, Tegenu M. Collaborative DTM reduces hospitalization and healthcare costs in patients with diabetes treated with polypharmacy. Am J Manag Care. 2014 Mar 1;20(3):e72-81. PMID 24773329
- [Background] Davidson MB. The effectiveness of nurse- and pharmacist-directed care in diabetes disease management: a narrative review. Curr Diabetes Rev. 2007 Nov;3(4):280-6. doi: 10.2174/157339907782330058. PMID 18220688
- [Background] Wubben DP, Vivian EM. Effects of pharmacist outpatient interventions on adults with diabetes mellitus: a systematic review. Pharmacotherapy. 2008 Apr;28(4):421-36. doi: 10.1592/phco.28.4.421. PMID 18363526
- [Background] Zullig LL, Melnyk SD, Stechuchak KM, McCant F, Danus S, Oddone E, Bastian L, Olsen M, Edelman D, Rakley S, Morey M, Bosworth HB. The Cardiovascular Intervention Improvement Telemedicine Study (CITIES): rationale for a tailored behavioral and educational pharmacist-administered intervention for achieving cardiovascular disease risk reduction. Telemed J E Health. 2014 Feb;20(2):135-43. doi: 10.1089/tmj.2013.0145. Epub 2013 Dec 4. PMID 24303930
- [Background] Maxwell LG, McFarland MS, Baker JW, Cassidy RF. Evaluation of the Impact of a Pharmacist-Led Telehealth Clinic on Diabetes-Related Goals of Therapy in a Veteran Population. Pharmacotherapy. 2016 Mar;36(3):348-56. doi: 10.1002/phar.1719. Epub 2016 Mar 11. PMID 26877253
- [Background] Littauer SL, Dixon DL, Mishra VK, Sisson EM, Salgado TM. Pharmacists providing care in the outpatient setting through telemedicine models: a narrative review. Pharm Pract (Granada). 2017 Oct-Dec;15(4):1134. doi: 10.18549/PharmPract.2017.04.1134. Epub 2017 Dec 19. PMID 29317927
- [Background] Barr PJ, McElnay JC, Hughes CM. Connected health care: the future of health care and the role of the pharmacist. J Eval Clin Pract. 2012 Feb;18(1):56-62. doi: 10.1111/j.1365-2753.2010.01522.x. Epub 2010 Aug 4. PMID 20698917
- [Background] Hughes JD, Wibowo Y, Sunderland B, Hoti K. The role of the pharmacist in the management of type 2 diabetes: current insights and future directions. Integr Pharm Res Pract. 2017 Jan 16;6:15-27. doi: 10.2147/IPRP.S103783. eCollection 2017. PMID 29354547
- [Background] Nye AM. A Clinical Pharmacist in Telehealth Team Care for Rural Patients with Diabetes. N C Med J. 2017 May-Jun;78(3):183-184. doi: 10.18043/ncm.78.3.183. No abstract available. PMID 28576957
- [Background] Emilia Romagna region. Causes of non-adherence to the diagnostic-therapeutic treatment of diabetes mellitus: a qualitative-quantitative study for improvement - Final report. June 2018

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment took place in the first 15 days of the operating period (November 1, 2018 - October 31, 2019). The patients were enrolled at the only experimentation center represented by La Regina pharmacy, a community pharmacy in a small rural center in southern Italy.
Pre-assignment Details: None of the enrolled patients were excluded from the ongoing trial. All patients completed the entire observation period.
Period: Overall Study
Arm/Group | Group Study
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Study participants were assigned the whole study group.
Groups:
- Group Study: Enrolled patients include people with reduced glucose tolerance, or impaired fasting blood sugar, or type 2 diabetes free of organ complications, or type 2 diabetes with chronic complications.
Arm/Group | Group Study
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (9.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Italy | 40

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Adherence to the PDTA
Description: Measure of the variation - compared to a historical cohort - of the percentage of adherence to PDTA (patients who performed the scheduled checks at 3-6-12 months / total of patients enrolled x 100) in the cohort of the patients enrolled in the study and therefore followed from a case manager identified in the community pharmacist with the opportunity to perform the checks provided in telemedicine and in self-analysis, thanks to the exploitation of "pharmacy of service".
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Groups:
- Group Study: The patients enrolled were 40.
  Based on the staging of diabetic disease, the enrolled population was made up as follows:
  * reduced glucose tolerance
  * impaired fasting blood sugar
  * type 2 diabetes free of organ complications
  * type 2 diabetes with chronic complications
Arm/Group | Group Study
Number analyzed (Participants) | 40
percentage of participants
  Percentage of adherence to PDTA - 3 months | 98
  Percentage of adherence to PDTA - 6 months | 98
  Percentage of adherence to PDTA - 12 months | 98

2. Secondary Outcome: Waiting Time
Description: variation in waiting times for the execution of the examinations envisaged by the PDTA - Difference of waiting times for the execution of diagnostic investigations between traditional model and experimental model (difference expressed in days)
Time Frame: 365 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group Study
Number analyzed (Participants) | 40
days
  Electrocardiogram waiting list | 117 (57.5)
  Fundus Oculi waiting list | 120 (50)

3. Secondary Outcome: Levels of Arterial Pressure
Description: variation of arterial pressure (Systolic, Diastolic) (mmHg)
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Group Study
Number analyzed (Participants) | 40
percentage of change
  Systolic pressure variation | -13 (12)
  Diastolic pressure variation | -9 (16)

4. Secondary Outcome: Levels of HbA1c
Description: variation of HbA1c levels (%) when the patient is followed by the community pharmacist as a case manager, as a result of greater adherence to therapy
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Group Study
Number analyzed (Participants) | 40
percentage of change | -4 (16)

5. Secondary Outcome: Levels of LDL-cholesterol
Description: variation of LDL-cholesterol (mg/dl) when the patient is followed by the community pharmacist as a case manager, as a result of greater adherence to therapy
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percentage of variation
Arm/Group | Group Study
Number analyzed (Participants) | 40
percentage of variation | -10 (27)

6. Secondary Outcome: Economic Impact
Description: Evaluation of the economic impact secondary to the establishment of the figure of the community pharmacist as Case Manager and to the use of the "pharmacy of service" (Comparison costs/benefits in euro between traditional assistence model and this innovative assistance model) ( comparison between the costs currently incurred by the Italian health care system for the assistance to patients with type 2 diabetes and the related benefits and costs deriving from the adoption of a care model such as the one object of research and the relative benefits)
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: euro/patient/year
Arm/Group | Group Study
Number analyzed (Participants) | 40
euro/patient/year | 210.25 (80.25)

ADVERSE EVENTS:
Time Frame: 12 months
Description: There wasn't any risk of adverse event.
Groups:
- Group Study: The 40 patients enrolled were 50% men and 50% women. The average age was 64.5 years. The median of the comorbidities presented by the participants was two, and in 33% (n = 13) of the cases there were more than 2 comorbidities per patient.
  Based on the staging of diabetic disease, the enrolled population was made up as follows:
  * reduced glucose tolerance 15%
  * impaired fasting blood sugar 5%
  * type 2 diabetes free of organ complications 38%
  * type 2 diabetes with chronic complications 42%
Arm/Group | Group Study
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group Study (N=40)
Description (Cardiac disorders) | 0 (0) — No significant adverse events were detected during the study
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group Study (N=40)
Not Serious Adverse Event (Cardiac disorders) | 0 (0) — No significant adverse events were detected during the study

LIMITATIONS AND CAVEATS:
The monocentric nature of the study and the small number of patients, however statistically adequate, they represent limits, which can be overcome with the replication of the study on more than one wide scale.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT03752567/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT03752567/ICF_001.pdf